CLINICAL TRIAL: NCT05693792
Title: A Six-Month Prospective Follow-Up Study of WB001 in Mild to Moderate Postpartum Depression
Brief Title: A Six-Month Prospective Follow-Up Study of WB001
Status: Withdrawn | Type: Observational
Why Stopped: Internal company decision
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Other Study IDs: WB001-002
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Postpartum Depression
Keywords: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Follow-up Group: Participants randomized to {WB001+TAU} and {ED001+TAU} in the parent study (WB001-001) will be assessed for 6 months following treatment completion.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No treatment regimen will be deployed in this follow-up study.

SUMMARY:
This study is a 6-month follow-up study to WB001-001 conducted to assess and evaluate the durability of the effect of {WB001+TAU} beyond the 8-week treatment period.

DETAILED DESCRIPTION:
This study is a 6-month prospective, observational follow-up study to the WB001-001 trial. Participants will be a convenience sample of those enrolled in the WB001-001 parent trial who consent to participate in a follow-up study at baseline for WB001-001. After completion of WB001-001's EOT assessment, those consenting to participate in the current study will be screened to confirm eligibility. Eligible participants will complete six assessment batteries (patient-reported outcomes [PROs]) on a monthly basis for a 6-month observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Must have prior enrollment in the WB001-001 trial and completion of Week 8/EOT
2. Must be willing and able to comply with all study procedures

Exclusion Criteria:

1. Documented AE or SAE at WB001-001 Week 8 related to participant safety, by Investigator judgement

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants in the current study will be a convenience sample of those enrolled in the WB001-001 parent trial who consent to participate in a follow-up study at baseline for WB001-001.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-06-08 (Estimated); Study Completion 2024-06-08 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Change from Baseline to Week 4; Change from Baseline to Week 8
  Clinician-rated measure of depression. The HAM-D6 is a subset of the HAM-D17 that assesses the 6 core items associated with major depression. Scores range from 0-22, where higher scores indicate greater depression severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Change from Baseline to Week 4; Change from Baseline to Week 8; Change from Baseline to Week 12; Change from Baseline to Week 16; Change from Baseline to Week 20; Change from Baseline to Week 24
  Measure of depression. A 9-item self-report questionnaire where total scores range from 0 to 27, with higher scores indicating greater levels of depression.
Edinburgh Postpartum Depression Scale (EPDS) | Change from Baseline to Week 4; Change from Baseline to Week 8; Change from Baseline to Week 12; Change from Baseline to Week 16; Change from Baseline to Week 20; Change from Baseline to Week 24
  Measure of postpartum depression. A 10-item self-report questionnaire that assesses depression criteria and yields a total score from 0 to 30 where higher scores denote greater depression.
Generalized Anxiety Disorder Questionnaire (GAD-7) | Change from Baseline to Week 4; Change from Baseline to Week 8; Change from Baseline to Week 12; Change from Baseline to Week 16; Change from Baseline to Week 20; Change from Baseline to Week 24
  Measure of anxiety. A 7-item brief self-report questionnaire, where total score range is between 0-21, with higher scores indicate greater levels of anxiety.
Mother-to-Infant Bonding Scale (MIBS) | Change from Baseline to Week 4; Change from Baseline to Week 8; Change from Baseline to Week 12; Change from Baseline to Week 16; Change from Baseline to Week 20; Change from Baseline to Week 24
  Measure of mother-infant bond. An 8-item self-report questionnaire, where total scores range from 0 to 24, with lower scores indicating good bonding.
Patient Global Impression scale (PGI) | Change from Baseline to Week 4; Change from Baseline to Week 8; Change from Baseline to Week 12; Change from Baseline to Week 16; Change from Baseline to Week 20; Change from Baseline to Week 24
  Measure of disease severity. A single-item scale asking respondents to rate the severity of their disease.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Change from Baseline to Week 4; Change from Baseline to Week 8; Change from Baseline to Week 12; Change from Baseline to Week 16; Change from Baseline to Week 20; Change from Baseline to Week 24
  Measure of risk for suicide. A clinician-administered assessment that measures four constructs: the severity of ideation, the intensity of ideation, behavior, and lethality. The C-SSRS consists of 10 categories with binary responses (Yes or No) to indicate the presence or absence of the behavior with a numerical score outcome.

REFERENCES:
- See also: [Study Evaluating the Efficacy and Safety of a Digital Therapeutic as an Adjunct to TAU in Postpartum Depression] — https://clinicaltrials.gov/ct2/show/NCT05551195